CLINICAL TRIAL: NCT05226104
Title: Investigating the Efficacy of a Fractionated 1927nm Laser for Diffuse Pigmentation and Actinic Changes
Brief Title: Fractionated 1927nm Laser for Diffuse Pigmentation and Actinic Changes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abby Culver, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-1191
Record Dates: First submitted 2022-01-10; First posted 2022-02-07 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Skin Pigment
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy Participants (Other): Subjects who are interested in treatment for facial fine lines and wrinkles will be recruited for the study.
  Interventions: Device: MOXI

INTERVENTIONS:
Device: MOXI — Patients will receive treatment using f1927 devices and will be treated twice over the affected areas, once each month for a total of two months.

SUMMARY:
This is a single-site, non-randomized, non-controlled study at UT Southwestern Medical Center at Dallas in the Department of Plastic Surgery designed to follow up to 30 qualified and consenting subjects receiving a fractionated 1927 combination treatments for diffuse hyperpigmentation and/or melasma. Patients will receive treatment using f1927 devices and will be treated twice over the affected areas, once each month for a total of two months, followed by two follow-up visits at 1-month and 3-months post-treatment.

DETAILED DESCRIPTION:
This is a prospective, non-controlled study where subjects will receive treatment using f1927 devices and will be treated twice over the affected areas of the face once each month for a total of two months. Patients will be evaluated at 1-month and 3-months post-treatment to monitor the clinical effects of treatment. Overall assessment of treatment efficacy will be based on evaluation of standard and close-up photography using pre- and post-procedural photos as well as images obtained by the Vectra H2 3D Imaging System. Baseline changes in the visualization and numeric analysis of pigmented areas will be evaluated utilizing the 3D Facial Skin Analysis software on the H2 System. Subjects will also undergo non-invasive skin measurements using optical coherence tomography (OCT) to noninvasively gather topographical and histological images of pre- and post-treated skin. Screening, treatment(s) with f1927, and OCT measurements are all for research purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults between 20-60 years of age.
2. Fitzpatrick skin type I-IV.
3. Individuals deemed by the Investigator to have a significant amount of pigmentation/melasma and that desire correction of this condition.
4. Individuals willing to withhold aesthetic therapies, or other therapies judged to potentially impact results to the treatment areas for the duration of the study.
5. Women of childbearing potential who agree to take a urine pregnancy test at the Screening visit or when deemed by Investigator. Women of childbearing potential must have a negative urine pregnancy test and must not be lactating at Screening. Women must be willing and able to use an acceptable method of birth control (see below) during the study. Women will not be considered of childbearing potential if one of the following is documented - postmenopausal for at least 12 months prior to study, without a uterus and/or both ovaries, bilateral tubal ligation at least 6 months prior to study enrollment
6. Individuals of childbearing potential who use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:

   * Established use of hormonal contraception (oral, injected, implanted, patch or vaginal ring)
   * Barrier methods with spermicide: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
   * Intrauterine device (IUD) or intrauterine system (IUS)
   * Surgical sterilization (e.g. vasectomy confirmed to be effective by sperm count check, tubal occlusion, hysterectomy, bilateral salpingectomy/oophorectomy)
   * Abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal methods are not acceptable forms of contraception
7. Individuals who can read, speak, write and understand English and who are willing to provide written informed consent.
8. Individuals willing to sign a photography release.
9. Individuals willing and able to cooperate with all study requirements for the duration of the study.

Exclusion Criteria:

1. Fitzpatrick skin type V-VI.
2. Known allergies to general skin care products.
3. Sensitivity to topical lidocaine or ester-based local anesthetics.
4. Active systemic or local conditions that may affect wound healing.
5. Current or recent history of inflammatory skin disease, infection or unhealed wound in the proposed treatment area(s).
6. History of systemic granulomatous diseases, either active or inactive, (e.g. Sarcoid, Wegener's, TB, etc.) or connective tissue diseases (e.g. lupus, dermatomyosistis, etc.).
7. Recent history of significant trauma to the areas to be treated (< 6 months).
8. Significant scarring, other than acne scars, in the area(s) to be treated.
9. Current or history of hypertrophic scarring or keloid scars.
10. Severe or cystic and clinically significant acne on the area(s) to be treated.
11. Tattoos in the area to be treated.
12. Observable suntan, nevi, excessive hair, etc. or other dermal conditions on the treatment area(s) of the face that might influence study results in the opinion of the Investigator.
13. Individuals who currently have cancerous or pre-cancerous lesions in the area(s) to be treated and/or with a history of skin cancer.
14. Individuals with skin pathology and/or pre-existing dermatologic condition in the treatment area (i.e. psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation) that the Investigator deems inappropriate for participation or could interfere with outcomes of the study.
15. History of chronic drug or alcohol use.
16. Microdermabrasion or glycolic acid treatment to the treatment area(s) within 4 weeks of study participation or who plan on having this treatment during the study.
17. History of the following cosmetic treatments in the area(s) to be treated:

    * Injectable filler of any type within the past 2 weeks
    * Neurotoxins within the past week
    * Ablative resurfacing laser treatment within the past 6 months
    * Non-ablative, rejuvenative laser or light treatment within the past 6 months
    * Chemical peel or dermabrasion within the past 3 months
18. Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study devices.
19. History of using the following prescription medications:

    * Accutane or other systemic retinoids within the past 6 months
    * Topical retinoids within the past 4 weeks
    * Prescription strength lightening devices (e.g. hydroquinone, tretinoin, AHA, BHA, poly-hydroxy acids, 4-hydroxyanisole alone or combined with tretinoin, etc.) within 4 months
    * Any anti-wrinkle or skin lightening devices, or topical or systemic medication known to affect skin aging or dyschromia (e.g. devices containing alpha/beta/polyhydroxy acids, Vitamin C, soy, Q-10, hydroquinone, systemic or licorice extract (topically), Tego ®, Cosmo C250, gigawhite, lemon juice extract (topically), embilica extract, etc.) within 2 weeks
    * Antiplatelet agents/anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use), and/or
    * Psychiatric drugs that, in the Investigator's opinion, would impair the subject from understanding protocol requirements or understanding and signing consent.
20. Individuals who are pregnant or nursing or those planning on becoming pregnant during the study according to self-report.
21. Immunocompromised individuals or those currently using immunosuppressive medications and/or radiation.
22. Individuals with uncontrolled disease such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Those with multiple health conditions may still be excluded from participation even if conditions are controlled.
23. Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures planned during the course of the study.
24. Individuals who, in the Investigator's opinion, have a history of poor cooperation, unreliability or noncompliance with medical treatment.
25. Individuals who are unable to understand instructions or give informed consent
26. Individuals who have physical or psychological conditions which, in the opinion of the Investigator, makes them unable to complete the study per protocol (e.g. not likely to avoid other cosmetic treatments to area; not likely to stay in study for entire duration due to other commitments; or those with concomitant conditions that may develop symptoms that might confuse or confound study treatments or assessments).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby Culver, MD, Principal Investigator — UT Southwestern; Jeffrey Kenkel, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Department of Plastic Surgery, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 patients underwent two treatments with non-ablative, f1927nm laser.
Groups:
- Non-ablative f1927nm Laser: Subjects who are interested in treatment for facial fine lines and wrinkles will be recruited for the study.
  MOXI: Patients will receive treatment using f1927 devices and will be treated twice over the affected areas, once each month for a total of two months.
Period: Overall Study
Arm/Group | Non-ablative f1927nm Laser
Started | 27
Completed | 24
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Non-ablative f1927nm Laser
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 4
  Unknown or Not Reported | 0
Fitzpatrick Skin Prototype [Count of Participants; unit: Participants] — Subjects with Fitzpatrick Type 1-4 were enrolled in this study.
  Type I always burns, never tans (palest; freckles) Type II usually burns, tans minimally (light colored but darker than fair) Type III sometimes mild burn, tans uniformly (golden honey or olive) Type IV burns minimally, always tans well (moderate brown)
  Participants
    Type 1 | 4
    Type 2 | 7
    Type 3 | 6
    Type 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Dyspigmentation Spots
Description: Numeric analysis of dyspigmentation (spots) will be analyzed using VISIA System.
  The change from baseline was calculated at Month 1 and Month 3. An increase in the absolute count would indicate improvement.
Time Frame: Baseline, Month 1 and Month 3
Population: The left and right side of each participant's face was analyzed separately resulting in an n of 48.
Measure: Median (Standard Deviation); unit: Dyspigmentation Spots
Units Other Than Participants: Location
Groups:
- Location: Left; Location: Right: Subjects who are interested in treatment for facial fine lines and wrinkles will be recruited for the study.
  MOXI: Patients will receive treatment using f1927 devices and will be treated twice over the affected areas, once each month for a total of two months.
Arm/Group | Location: Left | Location: Right
Number analyzed (Participants) | 24 | 24
Number analyzed (Location) | 24 | 24
Dyspigmentation Spots
  Baseline | 48.3 (12.1) | 46 (11.8)
  Month 1 | 42.2 (13.8) | 42.5 (10.9)
  Month 3 | 46.1 (13.1) | 42.9 (10.8)

2. Primary Outcome: Change in UV Spots
Description: Numeric analysis of lesions resulting from photodamage will be analyzed using VISIA System.
  The change from baseline was calculated at Month 1 and Month 3. An increase in the absolute count would indicate improvement.
Time Frame: Baseline, Month 1 and Month 3
Population: The left and right side of each participant's face was analyzed separately resulting in an n of 48.
Measure: Median (Standard Deviation); unit: UV Spots
Units Other Than Participants: Location
Arm/Group | Location: Left | Location: Right
Number analyzed (Participants) | 24 | 24
Number analyzed (Location) | 24 | 24
UV Spots
  Baseline | 29.4 (9.9) | 25.4 (9.3)
  Month 1 | 22.4 (10.1) | 21.6 (9.7)
  Month 3 | 25.8 (9.6) | 24.3 (10.8)

3. Primary Outcome: Change in Brown Spots
Description: Numeric analysis of lentigines and melasma will be analyzed using the VISIA system.
  The change from baseline was calculated at Month 1 and Month 3. An increase in the absolute count would indicate improvement.
Time Frame: Baseline, Month 1 and Month 3
Population: The left and right side of each participant's face was analyzed separately resulting in an n of 48.
Measure: Median (Standard Deviation); unit: Brown Spots
Units Other Than Participants: Location
Arm/Group | Location: Left | Location: Right
Number analyzed (Participants) | 24 | 24
Number analyzed (Location) | 24 | 24
Brown Spots
  Baseline | 62.5 (9.1) | 60.3 (10.8)
  Month 1 | 56.3 (8.8) | 57.1 (8.8)
  Month 3 | 59.1 (10.1) | 58.6 (9.1)

4. Primary Outcome: Physician's Global Assessment Scores (PGAS)- Right Face
Description: Clinician evaluators assessed the right side of each participants 1 and 3 month photographs to subjectively score clinical improvement.
  PGAS Score Description 0 Clear, except for possible residual discoloration, 100% improvement.
  1. Almost clear, very significant clearance, 90% improvement; only minor evidence of hyperpigmentation remains.
  2. Marked improvement, significant improvement, 75% improvement. Some disease evidence of hyperpigmentation remains.
  3. Moderate improvement, intermediate between slight and marked improvement; 50% improvement in appearance of hyperpigmentation
  4. Slight improvement, some improvement, 25% improvement; significant evidence of hyperpigmentation remains
  5. No improvement; hyperpigmented condition unchanged
  6. Worse; condition worse than at week 0
Time Frame: Month 1 and Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-ablative f1927nm Laser
Number analyzed (Participants) | 24
score on a scale
  1 Month | 3.45 (1.23)
  3 Month | 3.60 (1.35)

5. Primary Outcome: Physician's Global Assessment Scores (PGAS)- Left Face
Description: Clinician evaluators assessed the left side of each participants 1 and 3 month photographs to subjectively score clinical improvement.
  PGAS Score Description 0 Clear, except for possible residual discoloration, 100% improvement.
  1. Almost clear, very significant clearance, 90% improvement; only minor evidence of hyperpigmentation remains.
  2. Marked improvement, significant improvement, 75% improvement. Some disease evidence of hyperpigmentation remains.
  3. Moderate improvement, intermediate between slight and marked improvement; 50% improvement in appearance of hyperpigmentation
  4. Slight improvement, some improvement, 25% improvement; significant evidence of hyperpigmentation remains
  5. No improvement; hyperpigmented condition unchanged
  6. Worse; condition worse than at week 0
Time Frame: Month 1 and Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-ablative f1927nm Laser
Number analyzed (Participants) | 24
score on a scale
  Month 1 | 3.44 (1.15)
  Month 3 | 3.72 (1.32)

6. Primary Outcome: Physician's Global Assessment Score (PGAS)- Overall
Description: Clinician evaluators assessed 1 and 3 month photographs to subjectively score clinical overall improvement.
  PGAS Score Description 0 Clear, except for possible residual discoloration, 100% improvement.
  1. Almost clear, very significant clearance, 90% improvement; only minor evidence of hyperpigmentation remains.
  2. Marked improvement, significant improvement, 75% improvement. Some disease evidence of hyperpigmentation remains.
  3. Moderate improvement, intermediate between slight and marked improvement; 50% improvement in appearance of hyperpigmentation
  4. Slight improvement, some improvement, 25% improvement; significant evidence of hyperpigmentation remains
  5. No improvement; hyperpigmented condition unchanged
  6. Worse; condition worse than at week 0
Time Frame: Month 1 and Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-ablative f1927nm Laser
Number analyzed (Participants) | 24
score on a scale
  Month 1 | 3.44 (1.14)
  Month 3 | 3.66 (1.28)

ADVERSE EVENTS:
Time Frame: Data was collected within a 3 month period.
Arm/Group | Non-ablative f1927nm Laser
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-ablative f1927nm Laser (N=27)
sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT05226104/Prot_SAP_000.pdf